CLINICAL TRIAL: NCT06852248
Title: Ureteric Identification Using Indocyanine Green Dye Versus Conventional Ureteric Stenting to Reduce Post-operative Pain and Surgical Morbidity During Endometriosis Surgery: A Pilot Trial (ICE Trial)
Brief Title: Ureteric Identification Using Indocyanine Green Dye Versus Conventional Ureteric Stenting to Reduce Post-operative Pain and Surgical Morbidity During Endometriosis Surgery
Acronym: ICE
Status: Recruiting | Type: Observational
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: LPR 3359
Record Dates: First submitted 2025-02-18; First posted 2025-02-28 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Endometriosis; Deep Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Indocyanine Green; Coloring Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ureteric stenting: One group will have conventional ureteric stenting (temporary tubes placed in the ureters).
  Interventions: Procedure: Ureteric stenting
- Indocyanine green (ICG) dye: One group will receive indocyanine green (ICG) dye injected into the ureters to make them visible under a special light.
  Interventions: Procedure: Indocyanine green (ICG) dye

INTERVENTIONS:
Procedure: Ureteric stenting — The ICE trial is a pilot study involving two methods for identifying the ureters (tubes connecting the kidneys to the bladder) during endometriosis surgery. One group will have conventional ureteric stenting (temporary tubes placed in the ureters)
  Groups: Ureteric stenting
Procedure: Indocyanine green (ICG) dye — The ICE trial is a pilot study involving two methods for identifying the ureters (tubes connecting the kidneys to the bladder) during endometriosis surgery. One group will receive indocyanine green (ICG) dye injected into the ureters to make them visible under a special light.
  Groups: Indocyanine green (ICG) dye

SUMMARY:
Endometriosis is a common (around 1 in 10 women), non-cancerous condition where tissue similar to the womb lining is found growing elsewhere, most commonly inside the pelvis. Symptoms vary but can include intense pelvic pain and infertility.

Endometriosis that is very deep and painful may need surgery, which risks damage to the tubes that drain urine from the kidneys to the bladder (ureters). To reduce this risk, surgeons may put tiny plastic tubes called "stents" inside the ureters. These stents can stay for up-to 4 weeks following surgery but can cause severe pain and blood in the urine. Squirting a dye into the ureters, rather than using stents, may cause less pain for women after surgery whilst not making the removal of endometriosis worse, the operation take longer, or increasing the rates of complications (such as bleeding or damage to internal organs). Before a full clinical study can be run, the investigators need to understand whether this is possible, by doing a feasibility study

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 50 years
* Scheduled for laparoscopic or robotic-assisted surgical excision of deep endometriosis (DE) where ureteric stenting is planned.
* Willing and able to provide consent for participation in the study

Exclusion Criteria:

* Confirmed or suspected pregnancy at the time of enrolment.
* Suspicion or confirmation of malignancy.
* History of ureteric injury from prior surgery or trauma
* Medically unfit for surgery due to the following conditions:

  * Uncontrolled diabetes mellitus.
  * Severe Chronic Obstructive Pulmonary Disease (COPD).
  * Hypertrophic cardiomyopathy or significant cardiac conditions (e.g., recent myocardial infarction, aortic stenosis).
  * History of stroke or severe kyphoscoliosis.
  * Uncontrolled hypertension.
* Body mass index (BMI): BMI greater than 45

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with deep endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of eligible women | 24 months
  The number of eligible women across 2 UK sites that are suitable for trial recruitment
Proportion of eligible women agreeing to participate | 24 months
  Number of women who are eligible that then take part in the trial
Attrition rate in follow up process | 24 months
  Recording the percentage of people who drop out before the completion
Missing data in follow up process | 24 months
  Recording how much data is missing from the follow up data
Acceptability of the trial interventions and follow-up processes | 24 months
  Recording how acceptable surgeons find the trial interventions and follow up process.
Acceptability of the trial interventions and follow-up processes | 24 months
  Recording how acceptable participants find the trial interventions and follow up process. This will be done using a focus group
Reasons for declining participation or withdrawal after agreeing to participate | 24 months
  Recording the list of reasons people withdraw from the study or decline to take part

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, Staffordshire, United Kingdom